CLINICAL TRIAL: NCT03710837
Title: The Effect of Pain Education on Multidisciplinary Healthcare Students' Understanding of Chronic Pain, Clinical Recommendations and Attitudes Towards People With Chronic Pain: a Mixed-methods Randomised Controlled Trial
Brief Title: The Effect of Pain Education on Multidisciplinary Healthcare Students' Understanding of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Mrs Jagjit Mankelow, Principal Investigator, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 095/18
Record Dates: First submitted 2018-10-09; First posted 2018-10-18 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Education; Healthcare professional students
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Multi disciplinary randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant information is pseudonymised using student numbers only. As soon is data is generated data will be fully anonymised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education (Experimental): Intervention: Pain neuroscience education group. One-off, 70 minute duration session delivered by Dr Cormac Ryan.
  Interventions: Other: Pain neuroscience education
- Red flag education (Experimental): Intervention: Red flags education group. One-off 70 minute duration session delivered by Dr Cormac Ryan.
  Interventions: Other: Red flag education

INTERVENTIONS:
Other: Pain neuroscience education — Two different lectures covering essential clinical skills but one designed to explore the hypothesis
  Other Names: Red flag education
  Arms: Pain neuroscience education
Other: Red flag education — Two different lectures covering essential clinical skills but one designed to explore the hypothesis
  Other Names: Pain neuroscience education
  Arms: Red flag education

SUMMARY:
Chronic pain is the leading cause of disability worldwide affecting just under 28 million people in the UK. Chronic pain conditions require a biopsychosocial rather than a biomedical model of care. Biomedical management lacks evidence of effectiveness but also has the potential to exacerbate the condition by raising fears and anxiety about potential pathological abnormalities.

Healthcare professionals often hold negative beliefs about people with chronic pain and view the condition within a biomedical framework. These negative attitudes can be observed at the pre-registration training stage of the health professionals' career. Thus, the pre-registration phase is an important point where an individual's understanding of, and beliefs about, pain and people with pain may be shaped for the future. The need for improved and better education of healthcare professionals to support best practice for low back pain with the aim of integrating professionals' management of low back pain and fostering innovation in practice is well recognised. This study seeks to quantify the benefits of pain education in knowledge, attitudes and beliefs. The findings may encourage other pre-registration institutions to deliver pain education in a more directed way and simultaneously support the International Association for the Study of Pain's (IASP) proposed integration pain education into existing curriculum.

DETAILED DESCRIPTION:
In 2011 Briggs et al described pain education at undergraduate level for healthcare professionals as 'woefully inadequate'. Pain Neurophysiology Education (PNE) can improve undergraduates' pain understanding/management, however previous RCTs used single discipline groups and immediate follow-up. Investigation of the effectiveness of this education on students across the multi-professional team with medium-to-long-term follow-up will provide important new information on the generalisability of existing data and whether or not any changes in pain understanding/management are maintained over time.

This study aims to contribute to the development of neuromusculoskeletal physiotherapy by identifying whether or not this education, which aims to up skill healthcare professionals of the future, is effective and can change their behaviours in practice to enhance patient care in chronic pain management. PNE has been shown to be useful in patient care in conjunction with other treatment methods. If this intervention is successful in altering pain attitudes and knowledge in keeping with modern science then students may feel more confident and able to manage pain post qualification. The findings of this study will support or refute the addition of PNE into healthcare professional undergraduate programmes.

ELIGIBILITY:
Inclusion Criteria: No previous pain education

* Pre-registration student at Teesside University in one of following six disciplines: paramedics, occupational therapists, physiotherapists, midwifery, nursing, diagnostic radiography.

Exclusion Criteria: In depth previous pain education

* Disciplines other than those listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
HC-PAIRS questionnaire | 6 months
  Health Care Providers Pain and Impairment Relationship Scale - assessing attitudes and beliefs towards pain using a 13 item validated questionnaire. High score is a worse outcome. Scores range from 13-91.
Revised Neurophysiology Quiz | 6 months
  Measures knowledge of pain physiology using a 12 point validated questionnaire. Low score is poor sign. Scores range from 0-12.
Case vignette | 6 months
  Measures clinical practise behaviours in pain management. A validated proxy measure of clinical behaviour, MCQ weighted as appropriate or inappropriate according to current national clinical guidelines. A low score is good, and scores range from 4 to 20.
Red flag knowledge | 6 months
  Measures knowledge of red flags. Low score is a poor sign. Scores range from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martin, PhD, Study Director — Professor at Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No